CLINICAL TRIAL: NCT05005312
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL STUDY TO ASSESS THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-07321332 BOOSTED WITH RITONAVIR IN ADULT PARTICIPANTS WITH MODERATE HEPATIC IMPAIRMENT AND HEALTHY PARTICIPANTS WITH NORMAL HEPATIC FUNCTION
Brief Title: Study to Estimate the Effects of Hepatic Impairment on the Pharmacokinetics (PK) of PF-07321332
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C4671010
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Results first posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2022-10

CONDITIONS: Hepatic Impairment
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Healthy Volunteer
  Interventions: Drug: PF-07321332; Drug: Ritonavir
- Cohort 2 (Experimental): Hepatic Impairment
  Interventions: Drug: PF-07321332; Drug: Ritonavir

INTERVENTIONS:
Drug: PF-07321332 — Tablet
Drug: Ritonavir — PK Boosting agent

SUMMARY:
The study is to estimate the effect of hepatic impairment on the plasma PK of PF-07321332/ritonavir. Findings from this study will be used to develop dosing recommendations so that the dose and/or dosing interval may be adjusted appropriately in the presence of hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are classically healthy having no clinically relevant abnormalities. No known or suspected hepatic impairment
* Stable hepatic impairment that meets the criteria for Class B of the Child-Pugh Classification

Exclusion Criteria:

* Any condition possibly affecting drug absorption (eg, prior bariatric surgery, gastrectomy, ileal resection).
* Participants who have been vaccinated with COVID-19 vaccines within the past week of dosing
* A positive urine drug test, for illicit drugs, at Screening
* History of sensitivity reactions to ritonavir or any of the formulation components of PF-07321332 or ritonavir.
* eGFR <60 mL/min/1.73m2 based on the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) equation
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≥ upper limit of normal (ULN) (for healthy participants); AST or ALT > 5x ULN (for hepatic impairment participants)
* Albumin > ULN (for healthy participants);
* Prothrombin time > ULN (for healthy participants);
* Total bilirubin level ≥1.5 × ULN [NOTE: Participants with a history of Gilbert syndrome (and hence elevated total bilirubin) are eligible provided direct bilirubin level is ≤ ULN).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Orange County Research Center, Tustin, California
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671010

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventeen participants were assigned to treatment. One participant in the moderate hepatic impairment group was excluded from the safety and pharmacokinetic (PK) analysis set as this participant was randomized but was discontinued on Day 1 prior to dosing with study treatment PF-07321332. All 16 treated participants included 8 participants without hepatic impairment (Cohort 1) and 8 participants with moderate hepatic impairment (Cohort 2) completed the study.,
Groups:
- Normal Hepatic Function: Participants with normal hepatic function and matched, by average age, weight, and gender as much as practically possible with participants with moderate hepatic impairment. Participants received single 100 mg dose of PF-07321332 administered orally in combination with the PK boosting agent ritonavir administered as a 100 mg dose at -12, 0, 12, and 24 hours relative to PF-07321332 dosing.
- Moderate Hepatic Impairment: Moderate Hepatic Impairment: Participants with moderate hepatic impairment (grade B) with a Child-Pugh Score of 7-9. The CP classification assesses 5 hepatic parameters (serum total bilirubin, serum albumin, prothrombin time prolongation, ascites, and encephalopathy grade) on a scale of 1 to 3 (most severe derangement). Total moderate hepatic impairment score range is 7 to 9. Participants received single 100 mg dose of PF-07321332 administered orally in combination with the PK boosting agent ritonavir administered as a 100 mg dose at -12, 0, 12, and 24 hours relative to PF-07321332 dosing.
Period: Overall Study
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Started | 8 | 9
Treated | 8 | 8
Completed | 8 | 8 (One participant in the moderate hepatic impairment group was excluded from the safety and PK analysis set as this participant was randomized but was discontinued due to difficulty in venous access for blood draws on Day 1 prior to dosing with study treatment PF-07321332.)
Not Completed | 0 | 1
Not completed — Enrolled, but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.8 (6.16) | 56.1 (9.33) | 54.4 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 7 | 13
  Black or African American | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Plasma PF-07321332
Description: Cmax was the maximum observed plasma concentration and was directly observed from data. Concentration values below the lower limit of quantification (LLQ) were set to zero. Geometric mean analysis was on the log scale. Zero values were not included in geometric mean and geometric coefficient of variation calculation. The geometric coefficient of variation was expressed in percentage.
Time Frame: Day 1 at 0 (pre-dose for PF-07321332), 0.5, 1, 2, 3, 4, 6, 8, 10, and 12 hours, Day 2 at 24 and 36 hours, and Day 3 at 48 hours
Population: The PK parameter analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
micrograms per milliliter (ug/mL) | 1.886 (20) | 1.923 (48)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Test type: Other — The ratio and 90% CI were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 101.96, 90% CI 2-sided [74.20 to 140.11]

2. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of Plasma PF-07321332
Description: AUClast was area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration. The geometric coefficient of variation was expressed in percentage.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter/hour (ug*hr/mL)
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
micrograms/milliliter/hour (ug*hr/mL) | 14.97 (36) | 14.86 (43)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Test type: Other — The ratio and 90% CI were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 99.29, 90% CI 2-sided [70.81 to 139.21]

3. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Plasma PF-07321332
Description: AUCinf was defined as area under the plasma concentration-time curve from time zero to infinity. The geometric coefficient of variation was expressed in percentage.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*hr/mL
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
ug*hr/mL | 15.24 (36) | 15.06 (43)
Statistical Analysis 1: Comparison: Normal Hepatic Function vs Moderate Hepatic Impairment; Test type: Other — The ratio and 90% CI were expressed as percentages; ANOVA; Ratio of Adjusted Geometric Means = 98.78, 90% CI 2-sided [70.65 to 138.12]

4. Secondary Outcome: Number of Participants With an Treatment Emergent Adverse Event (TEAE)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent adverse event (TEAE) means event between first dose of study treatment and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. An SAE was an AE resulting in any of death; inpatient hospitalization; life-threatening experience; disability; congenital anomaly or deemed significant for any other reason.
Time Frame: Up to 2 months
Population: Population analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
Participants
  Participants with adverse events (All Causalities) | 3 | 4
  Participants with adverse events (Treatment Related) | 0 | 3

5. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs)
Description: ECG categorical summarization criteria: 1. PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): a) greater than or equal to (>=) 300 millisecond (msec), b) >=25% increase when baseline is > 200 msec or >=50% increase when baseline is less than or equal to (<=) 200 msec.
  2. QRS duration (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): a) >=140 msec, b) >=50% increase from baseline.
  3. QTcF interval (QT corrected using the Fridericia formula): a) >450 msec and <=480 msec, b) >480 msec and <=500 msec, c) >500 msec, d) >30 msec and <=60 msec increase from baseline, e) >60 msec increase from baseline.
Time Frame: Up to 2 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
Participants
  PR INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value ≥ 300 | 0 | 0
  PR INTERVAL NOT OTHERWISE SPECIFIED (MSEC): %Change ≥ 25/50% | 0 | 0
  QRS INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value ≥ 140 | 0 | 0
  QRS INTERVAL NOT OTHERWISE SPECIFIED (MSEC): %Change ≥ 50% | 0 | 0
  QT INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value > 500 | 0 | 0
  QTC INTERVAL NOT OTHERWISE SPECIFIED (MSEC): 450 < Value ≤ 480 | 0 | 0
  QTC INTERVAL NOT OTHERWISE SPECIFIED (MSEC): 480 < Value ≤ 500 | 0 | 0
  QTC INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Value > 500 | 0 | 0
  QTC INTERVAL NOT OTHERWISE SPECIFIED (MSEC): 30 < Change ≤ 60 | 0 | 0
  QTC INTERVAL NOT OTHERWISE SPECIFIED (MSEC): Change > 60 | 0 | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (MSEC): 450 < Value ≤ 480 | 0 | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (MSEC): 480 < Value ≤ 500 | 0 | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (MSEC): Value > 500 | 0 | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (MSEC): 30 < Change ≤ 60 | 0 | 0
  QTCF - FRIDERICIA'S CORRECTION FORMULA NOT OTHERWISE SPECIFIED (MSEC): Change > 60 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Vital Signs
Description: Criteria for vital signs abnormalities: increase or decrease from baseline in systolic blood pressure (SBP) >=30 mm Hg and increase or decrease from baseline in diastolic blood pressure (DBP) >=20 mm Hg; the value of SBP <90 mm Hg; the value of DBP <50 mm Hg; the value of pulse rate <40 bpm or >120 bpm.
Time Frame: Up to 2 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
Participants
  SBP: Value <90mmHg | 0 | 0
  SBP: Change >= 30 mmHg increase from baseline | 0 | 1
  SBP: Change >= 30 mmHg decrease from baseline | 0 | 0
  DBP: Value <50 mmHg | 0 | 0
  DBP: Change >= 20 mmHg increase from baseline | 0 | 0
  DBP: Change >= 20 mmHg decrease from baseline | 0 | 0
  Pulse Rate: Value <40 bpm | 0 | 0
  Pulse Rate: Value >120 bpm | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Laboratory Assessments (Without Regard to Baseline Abnormality)
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology; clinical chemistry; urinalysis.
Time Frame: Up to 2 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 8 | 8
Participants
  HEMATOLOGY: Platelets (10^3/mm^3) <0.5× lower limit of normal (LLN) | 0 | 1
  HEMATOLOGY: Eosinophils (10^3/mm^3) >1.2× upper limit of normal (ULN) | 1 | 2
  HEMATOLOGY: Monocytes (10^3/mm^3) >1.2× ULN | 0 | 1
  CLINICAL CHEMISTRY: Direct Bilirubin (mg/dL) >1.5× ULN: number analyzed (Participants) | 0 | 1
  CLINICAL CHEMISTRY: Direct Bilirubin (mg/dL) >1.5× ULN | 0 | 1
  CLINICAL CHEMISTRY: Aspartate Aminotransferase (U/L) >3.0× ULN | 0 | 1
  CLINICAL CHEMISTRY: Calcium (mg/dL) >1.1× ULN | 1 | 0
  CLINICAL CHEMISTRY: Glucose (mg/dL) >1.5× ULN | 0 | 1
  URINALYSIS: URINE Hemoglobin ≥1 | 1 | 0
  URINALYSIS: Urobilinogen ≥1 | 0 | 1
  URINALYSIS: Leukocyte Esterase ≥1 | 0 | 1
  URINALYSIS: Urine Microscopic Exam ≥1: number analyzed (Participants) | 1 | 0
  URINALYSIS: Urine Microscopic Exam ≥1 | 1 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment to the last dose of study treatment date +35 days (up to 2 months)
Description: The same event may appear as both an adverse event (AE) and an serious adverse event (SAE). An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Normal Hepatic Function | Moderate Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Hepatic Function (N=8) | Moderate Hepatic Impairment (N=8)
Nausea (Gastrointestinal disorders) | 0 | 1
Injection site pruritus (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT05005312/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT05005312/SAP_001.pdf